CLINICAL TRIAL: NCT01785368
Title: Implementing Referral Guidelines for Imaging Exams Requested Via the Emergency Department: Impact on Exam Relevance and Associated Delays
Brief Title: Referral Guidelines for Imaging Exams: Impact on Exam Relevance and Associated Delays
Acronym: RIU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LOCAL/2012/PR-01; 2013-A00113-42 (Other: ANSM)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Emergency Department Admission; Imaging Techniques
Keywords: guidelines; referral guidelines; exam delays; exam relevance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Before guideline implementation (Other): This study population consists of all patients for whom a participating ER doctor requests an imaging exam during the observation period BEFORE the implementation of the referral guidelines.
  [This study is composed of (1) a period of observation for 1 month BEFORE the implementation of the referral guidelines, followed by (2) the implementation of the referral guidelines, then (3) a 5-6 month washout period, and finally (4) a 1 month observational period AFTER the implementation of the referral guidelines.]
  Intervention: Baseline observation
  Interventions: Other: Baseline observation
- After guideline implementation (Other): This study population consists of all patients for whom a participating ER doctor requests an imaging exam during the observation period AFTER the implementation of the referral guideline.
  [This study is composed of (1) a period of observation for 1 month BEFORE the implementation of the referral guidelines, followed by (2) the implementation of the referral guidelines, then (3) a 5-6 month washout period, and finally (4) a 1 month observational period AFTER the implementation of the referral guidelines.]
  Intervention: Implementation of guidelines
  Interventions: Other: Implementation of guidelines

INTERVENTIONS:
Other: Implementation of guidelines — The participating ER doctors are required to request imaging exams for their patients according to a guide mutually constructed by the emergency and imaging departments of the Nîmes university hospital.
  Arms: After guideline implementation
Other: Baseline observation — During this period of the study, baseline data will be collected.
  Arms: Before guideline implementation

SUMMARY:
The main objective of this study is to evaluate the impact of the implementation of referral guidelines for imaging exams requested by the emergency department on exam relevance. The latter is assessed via the rate of suspected diagnoses that are confirmed by the requested exam.

DETAILED DESCRIPTION:
The secondary objectives of this study are to assess the impact of the implementation of referral guidelines for imaging exams requested by the emergency department on the following:

A. How exam results are classified in relation to the initial, suspected diagnosis.

B. Further aspects of exam relevance.

C. Delays associated with exams

D. Changes in practice in terms of type of examination, clinical situations, the number of tests ordered per patient, and emergency situations

E. Radiation and contrast agent exposures

ELIGIBILITY:
Inclusion Criteria:

* The patient (or his/her guardian/parent/person-of-trust) was correctly informed about the study
* A participating ER doctor has requested an imaging exam for the patient during one of the trial observation periods (ie the "before" period or the "after" period).

Exclusion Criteria:

* The patient is under judicial protection
* The patient (or his/her guardian/parent/person-of-trust) refuses to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8549 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06-02 (Actual); Study Completion 2014-06-02 (Actual)

PRIMARY OUTCOMES:
Change in the % of initial, suspected diagnoses that are confirmed positive by the requested exam | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.

SECONDARY OUTCOMES:
Change in the classification of exam results in relation to initial, suspected diagnosis | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Qualitative variable: (i) the suspected diagnosis is confirmed; (ii) the suspected diagnosis was not confirmed, the exam was normal; (iii) the suspected diagnosis was confirmed, and another unsuspected pathology was also found; (iv) the suspected diagnosis was not confirmed, and another unsuspected pathology was found.
  Measured over an observation period of 1 month.
Change in the % of requested exams that do not conform with the exam recommended by the implemented guidelines | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the positivity rate for each suspected diagnosis | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the % of exams performed identical to the exam requested | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the average delay between the time marked on the request and the exam. | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the average delay between the time marked on the request and the distribution of written exam results. | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the number of admissions in the emergency department | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the number of requests for imaging exams made by the emergency department | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the % of patients admitted to the emergency department and needing an imaging exam. | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the frequency of each type of exam carried out. | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the frequency of each type of clinical situation associated with imaging exams. | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the average number of imaging exams requested per patient | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the frequency of imaging exams requested per type of emergency situation | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  vital; imaging needed in 4 - 6 hours; imaging needed in 6 to 24h, scheduled for hospitalisation, external demand, social requirements
  Measured over an observation period of 1 month.
Change in the % agreement between the clinical situation coded by the emergency doctor and the radiologist | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the total radiation exposure per patient | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the frequency of injection of contrast agents | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.
Change in the frequency of patients requiring contrast agents AND whose exam results are classified as "the suspected diagnosis was not confirmed, exam normal" | baseline (days 0 to 30) versus the 6th month after implementation of guidelines
  Measured over an observation period of 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Richard, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Claret PG, Bobbia X, Macri F, Stowell A, Motte A, Landais P, Beregi JP, de La Coussaye JE. Impact of a computerized provider radiography order entry system without clinical decision support on emergency department medical imaging requests. Comput Methods Programs Biomed. 2016 Jun;129:82-8. doi: 10.1016/j.cmpb.2016.03.006. Epub 2016 Mar 17. PMID 27084323